CLINICAL TRIAL: NCT02498054
Title: Diabetic Mellitus Patients Glucose Range Awareness After Experiencing a New Blood Glucose Meter Feature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3135718
Record Dates: First submitted 2015-07-09; First posted 2015-07-15 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Education with new meter feature. (Experimental): Subjects experience a computer stimulation of a new meter feature ( colour range indicator) to help subjects interpret whether blood glucose results are low, in-range or high based on accepted guidance.
  Interventions: Behavioral: Education with new meter feature.

INTERVENTIONS:
Behavioral: Education with new meter feature. — The blood glucose meter has default settings for the colour range indicator which can be customized by the subjects and/or their healthcare professional. This colour range indicator will be presented to the subjects as a computer simulation to show subjects a range of typical blood glucose values and how this new feature would classify these results as being low (blue), in-range (green) or high (red).

SUMMARY:
A single visit & single arm study in 80 subjects with diabetes to determine if a short educational experience with a new blood glucose meter feature improves the ability of each subject to better classify glucose results into acceptable glucose ranges.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 1 diabetes Mellitus (T1DM) or Type 2 diabetes Mellitus (T2DM) for ≥ 3 months
* Currently performing self monitoring of blood glucose (SMBG) at home
* Aged ≥16 years

Exclusion Criteria:

* Previous use of any blood glucose meter with the colour range indicator feature to be evaluated in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Success rate to categorize blood glucose values into accepted ranges. | On average within 30 mins post intervention.

SECONDARY OUTCOMES:
Actual time taken to categorize blood glucose values into accepted ranges on the questionnaire provided. | On average within 30 mins post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Grady, Phd, Study Director — LifeScan
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom